CLINICAL TRIAL: NCT00401401
Title: An Open-labeled Trial With a Dose-escalation Part and a Parallel Group Design(1) Investigating Zalutumumab, an Anti-EGF Receptor Antibody, in Combination With Chemo-Radiation as First Line Treatment of Patients With Cancer of the Head and Neck (1) The Parallel Group Part Was Cancelled
Brief Title: Zalutumumab in Combination With Chemotherapy and Radiotherapy in Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: MTD was established and patients completed 16 months safety f-up and response assessments. It is considered of limited value to follow patients for 3 years.
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hx-EGFr-203
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-11

CONDITIONS: Head and Neck Cancer; Squamous Cell Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — zalutumumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Zalutumumab 4 mg/kg (Experimental): Zalutumumab 8 weekly infusions
  Interventions: Drug: zalutumumab; Drug: cisplatin; Procedure: Radiotherapy
- Zalutumumab 8 mg/kg (Experimental): Zalutumumab 8 weekly infusions
  Interventions: Drug: zalutumumab; Drug: cisplatin; Procedure: Radiotherapy
- Zalutumumab 12 mg/kg (Experimental): Zalutumumab 8 weekly infusions
  Interventions: Drug: zalutumumab; Drug: cisplatin; Procedure: Radiotherapy
- Zalutumumab 16 mg/kg (Experimental): Zalutumumab 8 weekly infusions
  Interventions: Drug: zalutumumab; Drug: cisplatin; Procedure: Radiotherapy

INTERVENTIONS:
Drug: zalutumumab — Eight weekly infusions
Drug: cisplatin — Infusions
Procedure: Radiotherapy — Daily in the treatment period

SUMMARY:
The purpose of this study is to investigate the safety of zalutumumab in combination with chemotherapy and radiotherapy as treatment of patients with head and neck cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with locoregionally advanced squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx

Exclusion Criteria:

* Prior treatment with radiotherapy in the head and neck area
* Prior treatment with chemotherapy
* Prior treatment with similar drugs (e.g. EGFr antibodies, EGFr inhibitors)
* Previous surgery with curative intent for head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gregoire, MD professor, Principal Investigator — St-Luc University Hospital, Brussels, Belgium
Locations (7):
- Oregon Health Sciences Center, Portland, Oregon, United States
- Belgium (2):
  - St-Luc University Hospital, Brussels
  - University Hospital Gasthuisberg, Leuven
- France (2):
  - Centre Georges-Francois Leclerc Hospital, Dijon
  - Hopital Bretonneau Clinique d'Oncologie et Radiothérapie, Tours
- Nijmegen University Hospital, Nijmegen, Netherlands
- Lund University Hospital, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Zalutumumab 8 mg/kg: Zalutumumab 8 weeky infusions
Period: Overall Study
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 12 mg/kg | Zalutumumab 16 mg/kg
Started | 6 | 6 | 6 | 12
Completed | 6 | 6 | 5 | 9
Not Completed | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 12 mg/kg | Zalutumumab 16 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 12 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Median (Full Range); unit: years] | 58 [46 to 64] | 54 [49 to 63] | 49 [22 to 60] | 52 [46 to 62] | 52 [22 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 1 | 7
  Male | 3 | 5 | 4 | 11 | 23
Region of Enrollment [Number; unit: participants]
  France | 0 | 0 | 1 | 3 | 4
  United States | 0 | 0 | 0 | 1 | 1
  Belgium | 4 | 4 | 3 | 6 | 17
  Sweden | 2 | 2 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of participants with at least one adverse event. All adverse events were collected during the 8 week treatment period and the following 4 weeks. Serious adverse events were collected during 3 years after the patient was allocated to the trial.
Time Frame: Overall Study
Measure: Number; unit: participants
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 12 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 12
participants | 6 | 6 | 6 | 12

2. Secondary Outcome: Overall Response
Description: Tumour response according to RECIST criteria J Natl Cancer Inst 2000;92:205-16 assessed by CT/MRI. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the longest diameter of target lesions; Overall Response (OR), CR+PR
Time Frame: Up to 3 years
Measure: Number; unit: Participants
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 12 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 12
Participants | 6 | 4 | 2 | 5

3. Secondary Outcome: Time to Response
Description: as for outcome 2
Time Frame: Up to 3 years
Population: Number of months between date of first infusion and date of best response
Measure: Median (Full Range); unit: months
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 12 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 6 | 4 | 2 | 5
months | 5.79 [3.8 to 12.0] | 3.98 [3.9 to 6.4] | 4.31 [4.2 to 4.5] | 5.80 [4.0 to 6.4]

4. Secondary Outcome: Best Overall Tumor Response
Description: as for outcome 2
Time Frame: Up to 3 years
Measure: Number; unit: Participants
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 12 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 12
Participants
  Complete response | 1 | 1 | 0 | 5
  Partial response | 5 | 3 | 2 | 0
  Stable disease | 0 | 2 | 2 | 6
  Progressive disease | 0 | 0 | 1 | 0
  Nonevaluable | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Zalutumumab 12 mg/kg | Zalutumumab 16 mg/kg
Serious Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 11/12
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 4 mg/kg (N=6) | Zalutumumab 8 mg/kg (N=6) | Zalutumumab 12 mg/kg (N=6) | Zalutumumab 16 mg/kg (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sigmoiditis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection in immunocompromised host (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Zalutumumab 4 mg/kg (N=6) | Zalutumumab 8 mg/kg (N=6) | Zalutumumab 12 mg/kg (N=6) | Zalutumumab 16 mg/kg (N=12)
Anaemia (Blood and lymphatic system disorders) | 3/3 (3) | 2 (3) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 6 (8) | 5 (6) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 5 (6) | 5 (6) | 9 (9)
Nausea (Gastrointestinal disorders) | 4 (9) | 5 (7) | 3 (5) | 6 (9)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (5) | 3 (3) | 6 (8)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Disease progression (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Fatigue (General disorders) | 5 (6) | 2 (2) | 1 (1) | 5 (5)
Mucosal inflammation (General disorders) | 6 (6) | 6 (7) | 5 (5) | 9 (9)
Pyrexia (General disorders) | 3 (4) | 2 (5) | 1 (1) | 2 (2)
Laryngitis (Infections and infestations) | 5 (5) | 6 (7) | 5 (6) | 9 (12)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Radiation skin injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (5) | 10 (13)
Weight decreased (Investigations) | 4 (4) | 2 (2) | 1 (1) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 2 (3) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 6 (7)

LIMITATIONS AND CAVEATS:
All adverse events were collected during the 8 week treatment period and for additional 4 weeks. Serious adverse events were collected for the extended follow-up period of up to 3 years.

The planned parallell group of the study was cancelled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site and the PI may be required to withhold the publication for up to 90 days. Subject to a reasoned request from the sponsor, the publication may be further delayed for a period up to 6 months from the date of first submission to the sponsor.

The sponsor has the right to require deletion of any trade secret, proprietary, or confidential information supplied by the sponsor to the site or the PI. The sponsor shall not otherwise have the right to censor publications.